CLINICAL TRIAL: NCT02155127
Title: Effects of a Walking Intervention in Older Patients With Chronic Kidney Disease: Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Patricia Painter, Associate Research Faculty, University of Utah
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB_00064407
Record Dates: First submitted 2014-06-02; First posted 2014-06-04 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Kidney Disease
Keywords: chronic kidney disease; physical function
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- walking intervention (Experimental): Subjects are randomized to walking/functional strength program with weekly coaching or usual care. The program is for 12 weeks. The intervention includes 3 lower extremity strengthening exercises, and progressive walking.
  Interventions: Behavioral: walking
- usual care (No Intervention): these subjects receive information on walking program, however do not receive any coaching over 12 weeks

INTERVENTIONS:
Behavioral: walking
  Arms: walking intervention

SUMMARY:
Chronic kidney disease (CKD) affects more than 26 million individuals (13 percent) of the U.S. population, with a projected 70 percent increase by the year 2015 to over 40 million individuals. Impairments in physical function and mobility limitations have been reported in older Chronic Kidney Disease patients, however the consequences of impaired functioning on participation in daily life and quality of life have not been studied. Early identification and interventions to mitigate deterioration in physical function and mobility should lead to improved health and quality of life outcomes in older patients with Chronic Kidney Disease. Although older individuals with Chronic Kidney Disease have reduced survival expectancy, maintaining physical function and mobility may contribute to longer active life expectancy, and higher quality of life despite their diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients over the age of 60 years
* Diagnosed with moderate to severe CKD (stage 2-4)
* Ambulatory (with or without use of an assistive device such as a cane or walker)
* Living in the community, cognitively able to provide consent and understand directions for the tests
* Cognitive ability to understand and carry out an independent home walking program
* Access and ability to communicate with study staff on a weekly basis and available for follow-up testing.

Exclusion Criteria:

* Inability to carry out a program of walking independently at home
* Unavailable for follow-up testing, estimated GFR >60 ml/minx1.73m2 and < 15 ml/minx1.73 m2
* Recent cardiac event (within the past 6 months)
* Uncontrolled hypertension
* Uncontrolled diabetes
* Pulmonary disease that may limit the ability to progress with walking
* Progressive neuromuscular disease
* Any orthopedic or neuromuscular condition that may be exacerbated by increased walking activity
* diabetic foot ulcer.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
walking speed | baseline to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Patricia L Painter, Ph.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States